CLINICAL TRIAL: NCT04010747
Title: Pilot Study of Motivational Interviewing for Loved Ones
Acronym: MILO-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H-41305; 5K23MH118373-04 (NIH); 2019P-000473 (Other: Beth Israel Deaconess Medical Center)
Record Dates: First submitted 2019-07-02; First posted 2019-07-08 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Psychotic Disorders; Psychosis; Psychotic Episode
Keywords: Parents; Family Members; Partner, Domestic
MeSH Terms: conditions — Psychotic Disorders | interventions — Motivational Interviewing; Waiting Lists

STUDY DESIGN:
Intervention Model Description: The first 30 participants to enroll in this study will receive a training intervention called "Motivational Interviewing for Loved Ones" (MILO).
  After that, participants will be randomly assigned to the intervention (MILO) or to a control condition involving a 30-minute mental health services consultation and a 6 week waitlist followed by the opportunity to participate in the MILO intervention ("Phase 2")
Who Masked: Outcomes Assessor
Masking Description: Prior to the crossover the study will be open label. After the crossover, the outcome assessor will be blinded to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing for Loved Ones (MILO) (Experimental): MILO consists of four sessions of "coaching" in communication skills called motivational interviewing. Participants meet with a trainer/therapist for each session. At the first session, participants learn about the ideas behind motivational interviewing. In the second session, participants practice motivational interviewing skills. In the third and fourth sessions, the participant and therapist discuss the participant's efforts to communicate with their loved one using MI skills. Participants will also be offered direct assistance with a referral to mental health treatment for their loved one.
  Interventions: Behavioral: Motivational Interviewing for Loved Ones (MILO)
- Mental Health Services Consultation and Waitlist (Active Comparator): This consultation will consist of a 30 minute appointment in which participants can speak with a clinician knowledgeable about psychosis treatment resources. He/she can recommend specific programs, educational websites, and/or support groups that might be relevant for the participant's family. Participants will then be placed on a 6-week waitlist, after which they will have the opportunity to participate in the active intervention (four sessions of MILO).
  Interventions: Behavioral: Motivational Interviewing for Loved Ones (MILO); Behavioral: Mental Health Services Consultation and Waitlist

INTERVENTIONS:
Behavioral: Motivational Interviewing for Loved Ones (MILO) — 4 sessions of behavioral coaching in motivational interviewing communication techniques
Behavioral: Mental Health Services Consultation and Waitlist — 1 session of individualized consultation on relevant mental health services for the IP and participating PCSO and 6 weeks on a waitlist, followed by opportunity to participate in MILO sessions.
  Arms: Mental Health Services Consultation and Waitlist

SUMMARY:
The study population for this research will include parents and concerned significant others (PCSO) of individuals experiencing recent (past five years) onset of a psychotic disorder (hereafter referred to as individuals with psychosis, "IP") who are not currently engaged with, or at risk for disengagement from, treatment. MILO is a brief and structured intervention that teaches motivational interviewing communication strategies. The initial aim (phase 1) of this pilot study is to evaluate feasibility of the intervention. The secondary aims are to evaluate the effectiveness of MILO for (1) enhancing the engagement of IP with evidence-based treatments and (2) reducing distress among PCSO. The investigators hypothesize that the intervention will be superior to control condition for both enhancing IP engagement with mental health services and reducing PCSO distress.

DETAILED DESCRIPTION:
First Episode Psychosis (FEP) often represents a time of crisis for young people and their families. Since peak onset occurs during late adolescence and early adulthood, the onset of serious mental health challenges can disrupt plans for education, relationships, and other milestones of independence. Although some psychoses are brief and self-limiting, more often these symptoms portend a potentially chronic and disabling psychiatric disorder such as schizophrenia. FEP can also be acutely dangerous: youth with FEP are far more likely to die in the year following their diagnosis relative to the general population of 16-30 year old's in the United States. Approximately 100,000 youth in the United States experience FEP every year. Young people identified by providers as experiencing FEP often slip through the cracks before they reach appropriate treatment. A review of privately insured adolescents and young adults in the US showed that 62% of young people in the US with FEP filled no outpatient prescriptions, and 41% received no outpatient psychotherapy, in the year following their index diagnosis. Among those who do have an initial encounter with specialized FEP outpatient care, high attrition is a common problem, with 30% of individuals initially enrolled in first episode programs dropping out prior to completing treatment.

Many individuals experiencing psychosis are reluctant to seek mental health treatment due to lack of insight and fear of psychiatric interventions. Young adults may be torn between distress and dissatisfaction relating to their symptoms and functioning, and mistrust of mental health providers and irritation with their parents' concern. Motivational Interviewing (MI) techniques are designed to elicit this ambivalence through nonjudgmental listening, so that discrepancies between current behaviors and ideal outcomes can be explored. Clinician-delivered MI has been identified as effective for enhancing adherence once individuals with psychosis are involved in care, and may also be useful for engaging those who are not yet interested in treatment. Several studies have found positive results in training and deploying non-professionals to use MI to influence others' health behaviors. MI training for parents and concerned significant others (PCSO) is a promising venue through which PCSO can specifically influence their loved one's decision to seek care and adhere to treatment plans.

MILO is a structured and goal oriented intervention that seeks to accomplish two aims. The primary aim is to facilitate the engagement of IP with evidence-based treatments. The secondary aim is to reduce the distress and increase the wellbeing of PCSO. The intervention will be trialed for feasibility (phase 1, n = 30) and then tested against a small "treatment as usual" (TAU) control arm (phase 2, n = 40). During phase 2, participants will be randomly assigned to either receive MILO (50%) or TAU (50%). The trial will involve a total of 70 participants.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Primary caregiver or other close contact of an individual within first 5 years of onset of a psychotic disorder who is poorly engaged or unengaged in psychiatric treatment

Exclusion Criteria:

* Not able to provide informed consent
* Not proficient in English
* History of developmental delay
* Current acute mental health problem or distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily R Kline, PhD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kline ER, Thibeau H, Sanders AS, English K, Davis BJ, Fenley AR, Keshavan MS. Motivational Interviewing for Loved Ones in Early Psychosis: Development and Pilot Feasibility Trial of a Brief Psychoeducational Intervention for Caregivers. Front Psychiatry. 2021 Apr 1;12:659568. doi: 10.3389/fpsyt.2021.659568. eCollection 2021. PMID 33868061
- See also: Website containing information for potential study participants (approved by BIDMC IRB) — http://milostudy.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivational Interviewing for Loved Ones (MILO) | Mental Health Services Consultation and Waitlist
Started | 53 | 18
Completed | 53 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing for Loved Ones (MILO) | Mental Health Services Consultation and Waitlist | Total
Number analyzed (Participants) | 53 | 18 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (8.5) | 60.1 (9.9) | 57.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 12 | 51
  Male | 14 | 6 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 3 | 7
  Black | 3 | 1 | 4
  Hispanic | 2 | 0 | 2
  White | 42 | 13 | 55
  Prefer not to state | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 18 | 71
Baseline mental health related appointments by the individual with psychosis (IP) in prior month [Mean (Standard Deviation); unit: number of appointments] — The participant will report the number of mental health related appointments attended by the IP during the past month via a structured survey. Population: Data are missing for 1 participant in the MILO group.
  number of appointments
    number analyzed (Participants) | 52 | 18 | 70
    (all) | 1.63 (1.62) | 2.00 (1.78) | 1.73 (1.66)
Baseline parents and concerned significant others (PCSO) expressed emotion [Mean (Standard Deviation); unit: score on a scale] — Caregiver attitudes toward individual with psychosis; measured via 20-item "family questionnaire" (FQ). The FQ has is a 20 item scale with a total score range of 20-80. Higher scores indicate more expressed emotion (i.e. critical and over-involved attitudes toward family member).
  score on a scale | 54.74 (8.42) | 54.83 (10.27) | 54.76 (8.85)
Baseline parents and concerned significant others (PCSO) distress [Mean (Standard Deviation); unit: score on a scale] — Symptoms of depression, anxiety, and behavioral disorders experienced by the PCSO; measured via the Perceived Stress Scale (PSS). The PSS is a 10 item questionnaire with a total score range of 0-40. Higher total scores indicate higher stress.
  score on a scale | 19.47 (5.75) | 19.50 (6.15) | 19.48 (5.81)
Baseline PCSO acquisition of motivational interviewing skills [Mean (Standard Deviation); unit: score on a scale] — PCSO will attempt to demonstrate motivational interviewing (MI) skills in a recorded role play; role play will be scored using a modified Motivational Interviewing Treatment Integrity Scale. Scores can range from 0 (poor MI skills demonstration) to 20 (expert MI skills demonstration). Higher scores represent increased proficiency in motivational interviewing skills: giving information, persuading with permission, questioning, reflecting, affirming, seeking collaboration, and emphasizing autonomy. Population: Data are missing for 2 participant in the MILO group.
  score on a scale
    number analyzed (Participants) | 51 | 18 | 69
    (all) | 10.98 (4.46) | 12.17 (5.44) | 11.29 (4.72)
Baseline PCSO beliefs and self confidence to parent [Mean (Standard Deviation); unit: score on a scale] — This outcome will be measured via the Parenting Self Agency Measure and only completed by those who identified as parents. The scale has 10 items rated by a 0% "Never"-100% "Always" slider scale. Higher scores rare associated with more parenting confidence. Population: Data are missing for 2 participant in the MILO group.
  score on a scale
    number analyzed (Participants) | 51 | 18 | 69
    (all) | 58.83 (11.99) | 55.21 (15.07) | 57.89 (12.85)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Mental Health Related Appointments Attended by the Individual With Psychosis (IP) in the Past 30 Days
Description: The participant will report the number of mental health related appointments attended by the IP during the past month via a structured survey.
Time Frame: Change from Baseline to 12 weeks
Population: There was missing data for 11 of the MILO and 1 of the Waitlist groups
Measure: Mean (Standard Deviation); unit: number of appointments
Arm/Group | Motivational Interviewing for Loved Ones (MILO) | Mental Health Services Consultation and Waitlist
Number analyzed (Participants) | 42 | 17
number of appointments | 0.29 (1.64) | -1.06 (1.95)

2. Secondary Outcome: Change in Parents and Concerned Significant Others (PCSO) Expressed Emotion
Description: Caregiver attitudes toward individual with psychosis; measured via 20-item "family questionnaire" (FQ). The FQ has is a 20 item scale with a total score range of 20-80. Higher scores indicate more expressed emotion (i.e. critical and over-involved attitudes toward family member).
Time Frame: Change from Baseline to 12 weeks
Population: There was missing data for 8 of the MILO and 1 of the Waitlist groups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Interviewing for Loved Ones (MILO) | Mental Health Services Consultation and Waitlist
Number analyzed (Participants) | 45 | 17
score on a scale | -7.82 (10.46) | -7.0 (11.24)

3. Secondary Outcome: Change in Parents and Concerned Significant Others (PCSO) Distress
Description: Symptoms of depression, anxiety, and behavioral disorders experienced by the PCSO; measured via the Perceived Stress Scale (PSS). The PSS is a 10 item questionnaire with a total score range of 0-40. Higher total scores indicate higher stress.
Time Frame: Change from Baseline to 12 weeks
Population: There was missing data for 8 of the MILO and 1 of the Waitlist groups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Interviewing for Loved Ones (MILO) | Mental Health Services Consultation and Waitlist
Number analyzed (Participants) | 45 | 17
score on a scale | -3.91 (5.86) | -4.47 (7.48)

4. Other Pre Specified Outcome: Change in Parents and Concerned Significant Others (PCSO) Acquisition of Motivational Interviewing Skills
Description: PCSO will attempt to demonstrate motivational interviewing (MI) skills in a recorded role play; role play will be scored using a modified Motivational Interviewing Treatment Integrity Scale. Scores can range from 0 (poor MI skills demonstration) to 20 (expert MI skills demonstration). Higher scores represent increased proficiency in motivational interviewing skills: giving information, persuading with permission, questioning, reflecting, affirming, seeking collaboration, and emphasizing autonomy.
Time Frame: Change from Baseline to 6 weeks
Population: There was missing data for 8 of the MILO and 4 of the Waitlist groups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Interviewing for Loved Ones (MILO) | Mental Health Services Consultation and Waitlist
Number analyzed (Participants) | 45 | 14
score on a scale | 5.09 (3.67) | 5.29 (4.41)

5. Other Pre Specified Outcome: Change in PCSO Beliefs and Self Confidence to Parent
Description: This outcome will be measured via the Parenting Self Agency Measure and only completed by those who identified as parents. The scale has 10 items rated by a 0% "Never"-100% "Always" slider scale. Higher scores rare associated with more parenting confidence.
Time Frame: Change from Baseline to 6 weeks
Population: There was missing data for 10 of the MILO and 1 of the Waitlist groups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Interviewing for Loved Ones (MILO) | Mental Health Services Consultation and Waitlist
Number analyzed (Participants) | 43 | 17
score on a scale | 5.59 (12.66) | 12.12 (13.13)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Motivational Interviewing for Loved Ones (MILO) | Mental Health Services Consultation and Waitlist
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/18
Other Adverse Events (participants affected / at risk) | 0/53 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/47/NCT04010747/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT04010747/ICF_000.pdf